CLINICAL TRIAL: NCT00451321
Title: TRX4 Therapeutic Evaluation of Different Multi-Dose Regimens in Type 1 Diabetes Mellitus (TTEDD)
Brief Title: TRX4 Monoclonal Antibody in Type 1 Diabetes (T1 DM)
Acronym: TTEDD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115493; TRX4005 (Other: Tolerx)
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: type 1 diabetes mellitus; diabetes mellitus type 1; type 1 diabetes; diabetes mellitus; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — otelixizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- otelixizumab (Experimental)
  Interventions: Drug: Otelixizumab

INTERVENTIONS:
Drug: Otelixizumab — Infusion

SUMMARY:
The purpose of this study is to optimize several multi-dose regimens of otelixizumab, determine the highest biologically active dose, evaluate biomarkers and surrogates of efficacy, and to evaluate the effects of each multi-dose regimen of otelixizumab against standard safety and efficacy parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adults 12 to 45 years old who are in good general health
* Confirmed diagnosis of insulin requiring type 1 diabetes mellitus with good glycemic control
* Measurable C-peptide levels

Exclusion Criteria:

* Females must not be pregnant or lactating and willing to practice contraception
* No prior malignancy, other than non-melanoma skin cancer
* Body Mass Index (BMI) > 32 at screening

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 88 (Actual)
Dates: Start 2006-07-31 (Actual); Primary Completion 2011-12-01 (Actual); Study Completion 2011-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- United States (16):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Pinellas Park, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Gulfport, Mississippi
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Mentor, Ohio
  - GSK Investigational Site, Rapid City, South Dakota
  - GSK Investigational Site, San Antonio, Texas
- GSK Investigational Site, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Keymeulen B, Vandemeulebroucke E, Ziegler AG, Mathieu C, Kaufman L, Hale G, Gorus F, Goldman M, Walter M, Candon S, Schandene L, Crenier L, De Block C, Seigneurin JM, De Pauw P, Pierard D, Weets I, Rebello P, Bird P, Berrie E, Frewin M, Waldmann H, Bach JF, Pipeleers D, Chatenoud L. Insulin needs after CD3-antibody therapy in new-onset type 1 diabetes. N Engl J Med. 2005 Jun 23;352(25):2598-608. doi: 10.1056/NEJMoa043980. PMID 15972866
- See also: Click here for more information on the TTEDD study — http://www.tolerx.com
- Available data/document: Statistical Analysis Plan: 115493 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115493 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115493 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115493 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115493 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115493 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115493 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 17 centers from United States and Canada during the period 31 July 2006 to 1 December 2011.
Pre-assignment Details: Participants from all 7 cohorts who had received a total dose <3.0 milligrams (mg) were analyzed as a separate treatment group. All other participants were analyzed according to the planned dose based on the cohort they belonged to.
Groups:
- Otelixizumab <3.0 mg: Participants from any of the 7 cohorts [3.1 mg, 3.1 mg (5 days), 4.35 mg, 4.35 mg (ITC-5), 4.35 mg (ITC-30), 6.85 mg and 8.85 mg] receiving a total Otelixizumab dose <3.0 mg during the study were analyzed in this cohort.
- Otelixizumab 3.1 mg: Participants in cohort 1 received one dose per day of Otelixizumab with doses 0.1 mg, 0.2 mg, 0.3 mg and then 0.5 mg x 5 as IV infusion administered over 2 hours for 8 consecutive days.
- Otelixizumab 3.1 mg (5 Days): Participants in cohort 5 received one dose per day of Otelixizumab with doses 0.2 mg, 0.4 mg, 0.6 mg, 0.8 mg and 1.1 mg as IV infusion administered over 30 minutes for 5 consecutive days.
- Otelixizumab 4.35 mg: Participants in cohort 2 received one dose per day of Otelixizumab with doses 0.1 mg, 0.2 mg, 0.3 mg, then 0.75 mg x 5 as IV infusion administered over 2 hours for 8 consecutive days.
- Otelixizumab 4.35 mg (ITC-15): Participants in ITC-15 cohort received one dose per day of Otelixizumab with doses 0.1 mg, 0.2 mg, 0.3 mg, then 0.75 x 5 as IV infusion administered over 15 minutes for 8 consecutive days.
- Otelixizumab 4.35 mg (ITC-30): Participants in ITC-30 cohort received one dose per day of Otelixizumab with doses 0.1 mg, 0.2 mg, 0.3 mg, then 0.75 x 5 as IV infusion administered over 30 minutes for 8 consecutive days.
- Otelixizumab 6.85 mg: Participants in cohort 3 received one dose per day of Otelixizumab with doses 0.1 mg, 0.2 mg, 0.3 mg, 0.75 mg, 1.0 mg, 1.25 mg, 1.5 mg and 1.75 mg as IV infusion administered over 2 hours for 8 consecutive days.
- Otelixizumab 8.85 mg: Participants in cohort 4 received one dose per day of Otelixizumab with doses 0.1 mg, 0.2 mg, 0.3 mg, 0.75 mg, 1.0 mg, 1.25 mg, 1.50 mg and 3.75 mg as IV infusion administered over 2 hours for 8 consecutive days.
Period: Overall Study
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Started | 8 | 15 | 18 | 19 | 7 | 9 | 6 | 6
Completed | 1 | 10 | 0 | 7 | 0 | 0 | 0 | 0
Not Completed | 7 | 5 | 18 | 12 | 7 | 9 | 6 | 6
Not completed — Lost to Follow-up | 3 | 3 | 1 | 3 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 4 | 0 | 0 | 0 | 0
Not completed — Study closed/terminated | 1 | 1 | 17 | 5 | 7 | 7 | 5 | 3
Not completed — Sponsor decision to amend protocol | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Participants from all 7 cohorts who had received a total dose <3.0 mg were analyzed as a separate treatment group. All other participants were analyzed according to the planned dose based on the cohort they belonged to.
Groups:
- Total: Total of all reporting groups
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg | Total
Number analyzed (Participants) | 8 | 15 | 18 | 19 | 7 | 9 | 6 | 6 | 88
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.8 (11.36) | 42.3 (13.25) | 18.9 (5.17) | 34.6 (9.89) | 36.1 (9.70) | 28.9 (10.74) | 37.2 (14.37) | 28.8 (6.79) | 31.6 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 5 | 9 | 4 | 5 | 3 | 2 | 39
  Male | 2 | 10 | 13 | 10 | 3 | 4 | 3 | 4 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 8 | 15 | 16 | 19 | 7 | 9 | 6 | 6 | 86
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE include adverse events that result in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Up to Month 24
Population: The 'All Subjects population' was defined as all participants who received at least one dose of study medication and was used in all study population and safety analyses. Participants from all 7 cohorts who had received a total dose <3.0 mg were analyzed as a separate treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Number analyzed (Participants) | 8 | 15 | 18 | 19 | 7 | 9 | 6 | 6
Participants
  Any AEs | 8 | 15 | 18 | 18 | 7 | 9 | 6 | 6
  Any SAEs | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 2

2. Primary Outcome: Number of Participants With Cytokine Release AE
Description: AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Cytokine release AEs were defined as occurring during dosing or within a limited time window after the last dose.
Time Frame: Up to Month 24
Population: All subjects Population. Participants from all 7 cohorts who had received a total dose <3.0 mg were analyzed as a separate treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Number analyzed (Participants) | 8 | 15 | 18 | 19 | 7 | 9 | 6 | 6
Participants | 8 | 11 | 18 | 17 | 7 | 9 | 6 | 6

3. Primary Outcome: Number of Participants With Abnormal Hematology Values of Potential Clinical Concern (PCC)
Description: Hematology parameters: hemoglobin, white blood cell (WBC) count, basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelet count, mean corpuscular volume, mean corpuscular hemoglobin, and mean corpuscular hemoglobin concentration were assessed for abnormal PCC values. Data for abnormal parameters (high and low) is presented. Only those parameters for which at least one value of PCC was reported are summarized.
Time Frame: Up to Month 48
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Number analyzed (Participants) | 8 | 15 | 18 | 19 | 7 | 9 | 6 | 6
Participants
  Lymphocytes, low | 4 | 12 | 18 | 17 | 7 | 9 | 5 | 5
  WBC, low | 3 | 4 | 12 | 5 | 3 | 5 | 3 | 4
  Hemoglobin, high | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils, low | 1 | 2 | 11 | 1 | 3 | 2 | 3 | 2
  Platelets, low | 0 | 2 | 4 | 2 | 0 | 0 | 0 | 0
  Platelets, high | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0

4. Primary Outcome: Number of Participants With Abnormal Clinical Chemistry Values of PCC
Description: Clinical chemistry parameters: alkaline phosphatase, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, gamma-glutamyl transferase, lactate dehydrogenase, lipids, blood urea nitrogen, creatinine, uric acid, sodium, potassium, chloride, carbon dioxide, creatinine phosphokinase, albumin, calcium, magnesium, glucose, phosphate, bicarbonate and total protein were assessed for abnormal PCC values. Data for abnormal parameters (high and low) is presented. Only those parameters for which at least one value of PCC was reported are summarized.
Time Frame: Up to Month 48
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Number analyzed (Participants) | 8 | 15 | 18 | 19 | 7 | 9 | 6 | 6
Participants
  ALT, high | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 0
  AST, high | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Fasting glucose, high | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Fasting glucose, low | 0 | 2 | 0 | 2 | 1 | 2 | 1 | 0
  Potassium, high | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bicarbonate, high | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Bicarbonate, low | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
  Calcium, low | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
  Magnesium, high | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase, high | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Total billirubin, high | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1

5. Primary Outcome: Number of Participants With Abnormal Urinalysis Dipstick Results
Description: Urinalysis parameters: Occult blood, Glucose urine, Ketones, Leukocyte esterase, Nitrite, pH, Protein urine were assessed. Abnormal values for occult blood and ketones were presented as 1+, 2+ and 3+ (the plus sign increases with a higher level of parameters: 1+=slightly positive, 2+=positive, 3+=high positive). Abnormal glucose urine values were presented as 50, 100, 250 and 1000 mg/dL. Abnormal nitrite values were presented as 'positive', and abnormal urine protein values were presented as 30 and 100 mg/dL.
Time Frame: Up to Month 48
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Number analyzed (Participants) | 8 | 15 | 18 | 19 | 7 | 9 | 6 | 6
Participants
  Occult blood, Day 8, 3+ | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Occult blood, Month 12, 1+ | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Occult blood, Month 12, 2+ | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0
  Occult blood, Month 12, 3+ | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Occult blood, Month 24, 1+ | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Occult blood, Month 24, 3+ | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Occult blood, Month 36, 2+ | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Occult blood, Month 36, 3+ | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Urine glucose, Day 8, 500 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Urine glucose, Month 12, 100 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Urine glucose, Month 12, 1000 | 2 | 5 | 0 | 5 | 1 | 2 | 0 | 2
  Urine glucose, Month 12, 250 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 1
  Urine glucose, Month 12, 50 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Urine glucose, Month 24, 100 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
  Urine glucose, Month 24, 1000 | 1 | 3 | 0 | 3 | 3 | 2 | 3 | 2
  Urine glucose, Month 24, 250 | 0 | 3 | 0 | 1 | 2 | 1 | 1 | 1
  Urine glucose, Month 24, 500 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1
  Urine glucose, Month 36, 1000 | 0 | 2 | 0 | 5 | 0 | 2 | 1 | 0
  Urine glucose, Month 36, 250 | 0 | 2 | 0 | 2 | 0 | 1 | 1 | 0
  Urine glucose, Month 36, 500 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Urine glucose, Month 48, 100 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Urine glucose, Month 48, 1000 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
  Urine glucose, Month 48, 250 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Urine ketones, Month 12, 1+ | 1 | 4 | 0 | 0 | 0 | 1 | 0 | 0
  Urine ketones, Month 12, 2+ | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0
  Urine ketones, Month 12, 3+ | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Urine ketones, Month 24, 1+ | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
  Urine ketones, Month 24, 2+ | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Urine ketones, Month 24, 3+ | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Urine ketones, Month 36, 1+ | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Urine ketones, Month 36, 2+ | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
  Urine ketones, Month 48, 1+ | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Leukocyte esterase, Month 12, 1+ | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Leukocyte esterase, Month 12, 2+ | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocyte esterase, Month 24, 1+ | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
  Leukocyte esterase, Month 24, 3+ | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Leukocyte esterase, Month 36, 1+ | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Nitrite, Month 12, positive | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Nitrite, Month 24, positive | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Nitrite, Month 36, positive | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Protein urine, Month 12, 30 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Protein urine, Month 24, 100 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Protein urine, Month 48, 30 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

6. Primary Outcome: Mean Overall Maximum Cytokines Level
Description: Levels of cytokines: interferon (IFN)-gamma, interleukin (IL)-10, IL-6 and tumor necrosis factor (TNF)-alpha were assessed. One sample was collected at Baseline, on dose Day 1 at 1, 2, 3, and 8 hours post-end of infusion (EOI) and on all other dosing days at pre-dose, and 1, 2, 3, and 8 hour post-EOI. After the completion of dosing, on Day 21 and Week 8, only the IL-10 level was assessed in the cytokine blood sample.
Time Frame: Up to Week 8
Population: All subjects Population. Only those participants available for analysis for the particular parameter are presented. Participants from all 7 cohorts who had received a total dose <3.0 mg were analyzed as a separate treatment group.
Measure: Mean (Standard Deviation); unit: Picograms per milliliter (pg/mL)
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Number analyzed (Participants) | 8 | 15 | 18 | 19 | 7 | 9 | 6 | 6
Picograms per milliliter (pg/mL)
  IFN-Gamma: number analyzed (Participants) | 1 | 1 | 4 | 3 | 1 | 1 | 2 | 3
  IFN-Gamma | 55.180 (NA) — Only one participant was analyzed, hence no data. | 20.170 (NA) — Only one participant was analyzed, hence no data. | 25.878 (19.0272) | 20.410 (15.6070) | 40.860 (NA) — Only one participant was analyzed, hence no data. | 9.730 (NA) — Only one participant was analyzed, hence no data. | 23.210 (12.7279) | 30.463 (23.4652)
  IL-10 | 146.084 (337.2007) | 44.609 (48.1712) | 58.743 (59.6380) | 75.879 (66.3559) | 80.267 (51.6266) | 82.786 (68.4322) | 193.065 (225.7715) | 82.547 (55.4185)
  IL-6 | 101.161 (193.9999) | 71.748 (78.0909) | 75.954 (63.2599) | 83.739 (65.1953) | 111.567 (115.1136) | 121.862 (99.0309) | 358.890 (544.0678) | 186.593 (200.7019)
  TNF-Alpha: number analyzed (Participants) | 8 | 15 | 17 | 19 | 7 | 9 | 6 | 6
  TNF-Alpha | 18.079 (10.2902) | 23.071 (29.9426) | 34.814 (40.1511) | 27.225 (37.5837) | 51.503 (36.9749) | 69.678 (145.2403) | 50.877 (74.6931) | 44.232 (51.2616)

7. Primary Outcome: Number of Participants With Positive Epstein Barr Virus (EBV) Viral Load
Description: EBV load was measured using quantitative polymerase chain reaction (PCR) method. If a participant had an EBV viral load of >100,000 copies/10^6 peripheral blood mononuclear cells (c/10^6 PBMC) lymphocytes at any time post-dose, the test was repeated immediately. Data for participants with abnormal viral load is presented.
Time Frame: Up to Month 18
Population: All subjects Population. Only those participants available at the specified time points were analyzed. Participants from all 7 cohorts who had received a total dose <3.0 mg were analyzed as a separate treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Number analyzed (Participants) | 8 | 15 | 18 | 19 | 7 | 9 | 6 | 6
Participants
  Screening, 1-10000: number analyzed (Participants) | 8 | 10 | 18 | 19 | 7 | 9 | 6 | 6
  Screening, 1-10000 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0
  Day 14, 1-10000: number analyzed (Participants) | 7 | 14 | 18 | 19 | 7 | 8 | 6 | 5
  Day 14, 1-10000 | 1 | 4 | 5 | 3 | 1 | 2 | 0 | 2
  Day 21, 1-10000: number analyzed (Participants) | 7 | 15 | 17 | 18 | 7 | 9 | 6 | 6
  Day 21, 1-10000 | 0 | 6 | 4 | 3 | 3 | 3 | 1 | 2
  Day 21, >10000: number analyzed (Participants) | 7 | 15 | 17 | 18 | 7 | 9 | 6 | 6
  Day 21, >10000 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 28, 1-10000: number analyzed (Participants) | 7 | 15 | 18 | 18 | 6 | 8 | 6 | 6
  Day 28, 1-10000 | 2 | 3 | 6 | 1 | 3 | 0 | 2 | 2
  Week 6, 1-10000: number analyzed (Participants) | 7 | 14 | 18 | 17 | 7 | 9 | 6 | 5
  Week 6, 1-10000 | 1 | 3 | 1 | 2 | 0 | 2 | 0 | 1
  Week 12, 1-10000: number analyzed (Participants) | 8 | 15 | 18 | 19 | 7 | 8 | 6 | 6
  Week 12, 1-10000 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Month 6, 1-10000: number analyzed (Participants) | 4 | 14 | 17 | 19 | 7 | 8 | 6 | 6
  Month 6, 1-10000 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Month 18, 1-10000: number analyzed (Participants) | 3 | 10 | 5 | 15 | 6 | 8 | 6 | 5
  Month 18, 1-10000 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 0
  Month 12, 1-10000: number analyzed (Participants) | 4 | 10 | 13 | 19 | 6 | 8 | 6 | 6
  Month 12, 1-10000 | 1 | 1 | 0 | 2 | 1 | 4 | 0 | 0

8. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration (AUClast) of Otelixizumab
Description: Pharmacokinetic (PK) samples were obtained at Baseline, and on all dose days except the final dose day, at pre-dose, EOI, and 4 hour post-SOI. On Dose Day 5, samples were collected at pre-dose, EOI, and 3.5, 4, 5, and 8-10 hour post-SOI. The lower limit of quantification was 0.019 micrograms per milliliter (µg/mL). The 'PK summary Population' was defined as participants in the 'All Subjects' Population for whom a pharmacokinetic sample was obtained and analyzed, and who received the full scheduled dose, as specified in the protocol. Only those participants available at the specified time points were analyzed.
Time Frame: At Baseline, and on all dose days except the final dose day, at pre-dose, EOI, and 4 hour post-start of infusion (SOI). On Dose Day 5, at pre-dose, EOI, and 3.5, 4, 5, and 8-10 hour post-SOI.
Population: PK summary Population. A limited comparison of the PK of free serum otelixizumab in adolescents and adults was attempted using the cumulative 3.1 mg dose regimen. However, there were insufficient quantifiable concentrations obtained in either group to allow meaningful conclusions to be drawn. Data for only quantifiable concentration is presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*micrograms per milliliter
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Number analyzed (Participants) | 0 | 14 | 0 | 15 | 7 | 9 | 6 | 3
Hour*micrograms per milliliter
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
  Day 1 |  |  |  | 0.03961 (139.9399) | 0.89984 (NA) — Only one participant was analyzed. |  |  |
  Day 4: number analyzed (Participants) | 0 | 2 | 0 | 12 | 3 | 1 | 4 | 2
  Day 4 |  | 0.01791 (48.7376) |  | 0.02752 (78.0203) | 0.06047 (809.8761) | 0.02595 (NA) — Only one participant was analyzed. | 0.01701 (47.9050) | 0.01370 (3.6149)
  Day 7: number analyzed (Participants) | 0 | 9 | 0 | 13 | 4 | 3 | 6 | 2
  Day 7 |  | 0.01789 (66.5077) |  | 0.08946 (161.9423) | 0.15744 (1108.625) | 0.02332 (27.3059) | 0.19563 (665.7708) | 0.20039 (80.3599)
  Day 8: number analyzed (Participants) | 0 | 10 | 0 | 13 | 4 | 6 | 6 | 3
  Day 8 |  | 0.01848 (73.4326) |  | 0.14250 (93.2214) | 0.08367 (280.2741) | 0.06685 (188.0044) | 0.62938 (256.4433) | 1.34488 (567.3411)

9. Secondary Outcome: Maximum Plasma Drug Concentration (Cmax) of Otelixizumab
Description: PK samples were obtained at Baseline, and on all dose days except the final dose day, at pre-dose, EOI, and 4 hour post-SOI. On Dose Day 5, samples were collected at pre-dose, EOI, and 3.5, 4, 5, and 8-10 hour post-SOI. The lower limit of quantification was 0.019 µg/mL. Only those participants available at the specified time points were analyzed.
Time Frame: At Baseline, and on all dose days except the final dose day, at pre-dose, EOI, and 4 hour post-SOI. On Dose Day 5, at pre-dose, EOI, and 3.5, 4, 5, and 8-10 hour post-SOI.
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Number analyzed (Participants) | 0 | 14 | 0 | 15 | 7 | 9 | 6 | 3
µg/mL
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
  Day 1 |  |  |  | 0.04399 (124.5265) | 0.06370 (NA) — Only one participant was analyzed. |  |  |
  Day 4: number analyzed (Participants) | 0 | 2 | 0 | 12 | 3 | 1 | 4 | 2
  Day 4 |  | 0.03050 (42.9529) |  | 0.03862 (41.1649) | 0.03041 (30.4698) | 0.03460 (NA) — Only one participant was analyzed. | 0.03160 (39.9688) | 0.02739 (3.6149)
  Day 7: number analyzed (Participants) | 0 | 9 | 0 | 13 | 4 | 3 | 6 | 2
  Day 7 |  | 0.02660 (37.1463) |  | 0.06715 (41.7413) | 0.05054 (41.4392) | 0.03075 (26.2309) | 0.12211 (118.6807) | 0.12601 (68.8972)
  Day 8: number analyzed (Participants) | 0 | 10 | 0 | 13 | 4 | 6 | 6 | 3
  Day 8 |  | 0.02988 (41.3271) |  | 0.06455 (45.7850) | 0.05519 (77.5056) | 0.03773 (41.5855) | 0.15106 (122.2439) | 0.23138 (254.9093)

10. Secondary Outcome: Time of Last Quantifiable Drug Concentration (Tlast) and Time of Occurrence of Maximum Plasma Drug Concentration (Tmax) of Otelixizumab
Description: PK samples were obtained at Baseline, and on all dose days except the final dose day, at pre-dose, EOI, and 4 hour SOI. On Dose Day 5, samples were collected at pre-dose, EOI, and 3.5, 4, 5, and 8-10 hour post-SOI. The lower limit of quantification was 0.019 µg/mL. Only those participants available at the specified time points were analyzed.
Time Frame: as for outcome 9
Population: as for outcome 8
Measure: Median (Full Range); unit: hour
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Number analyzed (Participants) | 0 | 14 | 0 | 15 | 7 | 9 | 6 | 3
hour
  tlast, Day 1: number analyzed (Participants) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
  tlast, Day 1 |  |  |  | 2.150 [2.08 to 4.05] | 22.250 [22.25 to 22.25] |  |  |
  tlast, Day 4: number analyzed (Participants) | 0 | 2 | 0 | 12 | 3 | 1 | 4 | 2
  tlast, Day 4 |  | 2.175 [2.13 to 2.22] |  | 2.133 [2.03 to 4.58] | 2.250 [2.25 to 23.58] | 2.500 [2.50 to 2.50] | 2.075 [2.00 to 2.17] | 2.000 [2.00 to 2.00]
  tlast, Day 7: number analyzed (Participants) | 0 | 9 | 0 | 13 | 4 | 3 | 6 | 2
  tlast, Day 7 |  | 2.217 [2.00 to 4.00] |  | 4.000 [2.00 to 23.67] | 12.375 [2.25 to 23.47] | 2.517 [2.50 to 2.53] | 4.000 [2.00 to 20.70] | 4.000 [4.00 to 4.00]
  tlast, Day 8: number analyzed (Participants) | 0 | 10 | 0 | 13 | 4 | 6 | 6 | 3
  tlast, Day 8 |  | 2.075 [2.00 to 4.00] |  | 5.033 [2.00 to 10.00] | 3.250 [1.75 to 8.32] | 3.500 [2.00 to 8.53] | 10.000 [4.03 to 10.17] | 12.000 [6.00 to 12.03]
  tmax, Day 1: number analyzed (Participants) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
  tmax, Day 1 |  |  |  | 2.083 [2.00 to 2.15] | 2.42 [2.42 to 2.42] |  |  |
  tmax, Day 4: number analyzed (Participants) | 0 | 2 | 0 | 12 | 3 | 1 | 4 | 2
  tmax, Day 4 |  | 2.175 [2.13 to 2.22] |  | 2.108 [1.92 to 2.53] | 2.250 [2.25 to 2.30] | 2.500 [2.50 to 2.50] | 2.075 [2.00 to 2.17] | 2.000 [2.00 to 2.00]
  tmax, Day 7: number analyzed (Participants) | 0 | 9 | 0 | 13 | 4 | 3 | 6 | 2
  tmax, Day 7 |  | 2.100 [2.00 to 2.33] |  | 2.083 [2.00 to 2.20] | 2.308 [2.25 to 22.47] | 2.517 [2.50 to 2.53] | 2.033 [2.00 to 2.33] | 3.042 [2.08 to 4.00]
  tmax, Day 8: number analyzed (Participants) | 0 | 10 | 0 | 13 | 4 | 6 | 6 | 3
  tmax, Day 8 |  | 2.075 [2.00 to 2.27] |  | 2.167 [2.00 to 2.75] | 2.000 [1.75 to 3.28] | 2.000 [2.00 to 2.50] | 3.500 [2.00 to 4.12] | 4.000 [4.00 to 4.03]

11. Secondary Outcome: Mean Lymphocytes Subsets (CD19+ B Cells, CD4+CD25hiFoxP3+ T Cells, CD8+CD25+FoxP3+ T Cells) Count
Description: One sample was collected at the screening visit and at Baseline. On dose Day 1, samples were collected at EOI and 4 hour post-SOI. On all other dosing days, samples were collected at pre-dose, EOI and 4 hour post-SOI. To obtain absolute counts for each lymphocyte subset (CD19+ B cells, CD4+CD25hiFoxP3+ T cells, CD8+CD25+FoxP3+ T cells) the proportion of total lymphocytes constituting that subset was multiplied by the total count for the same participant at the same time point. The data was collected on Baseline, Days 1 to 8, Days 14, 21, 28, Weeks 6, 8, 10, 12, Months 4, 5, 6, 12, 24, 36 and 48. However data for Days 8 and 28 is presented. The 'Pharmacodynamic (PD) summary population' was defined as participants in the 'All Subjects' Population for whom a PD sample was obtained and analyzed and who received the full scheduled dose, as specified in the protocol.
Time Frame: Day 8 and 28
Population: Only those participants available at the specified time points were analyzed. Data for only quantifiable concentration is presented.
Measure: Mean (Standard Deviation); unit: Cells per microliter
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Number analyzed (Participants) | 0 | 14 | 0 | 18 | 7 | 9 | 6 | 4
Cells per microliter
  CD19+ B Cells, Baseline: number analyzed (Participants) | 0 | 12 | 0 | 17 | 6 | 8 | 6 | 4
  CD19+ B Cells, Baseline |  | 0.187 (0.1360) |  | 0.247 (0.1029) | 0.288 (0.1173) | 0.393 (0.2125) | 0.200 (0.0873) | 0.220 (0.0922)
  CD19+ B Cells, Day 8, pre-dose |  | 0.182 (0.1697) |  | 0.180 (0.0627) | 0.146 (0.0305) | 0.203 (0.1019) | 0.099 (0.0468) | 0.151 (0.0906)
  CD19+ B Cells, Day 8, 15 minutes: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0
  CD19+ B Cells, Day 8, 15 minutes |  |  |  |  | 0.170 (0.0446) |  |  |
  CD19+ B Cells, Day 8, 30 minutes: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
  CD19+ B Cells, Day 8, 30 minutes |  |  |  |  |  | 0.204 (0.1094) |  |
  CD19+ B Cells, Day 8, 2 hours: number analyzed (Participants) | 0 | 14 | 0 | 17 | 0 | 0 | 6 | 4
  CD19+ B Cells, Day 8, 2 hours |  | 0.177 (0.1528) |  | 0.162 (0.0570) |  |  | 0.087 (0.0604) | 0.099 (0.0869)
  CD19+ B Cells, Day 8, 2.25 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0
  CD19+ B Cells, Day 8, 2.25 hours |  |  |  |  | 0.156 (0.0602) |  |  |
  CD19+ B Cells, Day 8, 2.5 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0
  CD19+ B Cells, Day 8, 2.5 hours |  |  |  |  |  | 0.161 (0.0737) |  |
  CD19+ B Cells, Day 8, 4 hours: number analyzed (Participants) | 0 | 13 | 0 | 17 | 0 | 0 | 6 | 4
  CD19+ B Cells, Day 8, 4 hours |  | 0.186 (0.1314) |  | 0.167 (0.0699) |  |  | 0.084 (0.0523) | 0.083 (0.0465)
  CD19+ B Cells, Day 28: number analyzed (Participants) | 0 | 14 | 0 | 16 | 6 | 8 | 6 | 4
  CD19+ B Cells, Day 28 |  | 0.198 (0.1978) |  | 0.210 (0.0634) | 0.156 (0.0553) | 0.279 (0.1558) | 0.167 (0.0470) | 0.153 (0.0783)
  CD4+CD25hiFoxP3+T cells, Baseline: number analyzed (Participants) | 0 | 12 | 0 | 18 | 6 | 8 | 6 | 4
  CD4+CD25hiFoxP3+T cells, Baseline |  | 0.0138 (0.01010) |  | 0.0099 (0.01142) | 0.0180 (0.00865) | 0.0165 (0.01262) | 0.0089 (0.00948) | 0.0379 (0.02839)
  CD4+CD25hiFoxP3+T cells, Day 8, pre-dose |  | 0.0062 (0.00497) |  | 0.0039 (0.00425) | 0.0056 (0.00488) | 0.0105 (0.00693) | 0.0028 (0.00180) | 0.0237 (0.01067)
  CD4+CD25hiFoxP3+T cells, Day 8, 15 minutes: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0
  CD4+CD25hiFoxP3+T cells, Day 8, 15 minutes |  |  |  |  | 0.0039 (0.00549) |  |  |
  CD4+CD25hiFoxP3+T cells, Day 8, 30 minutes: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
  CD4+CD25hiFoxP3+T cells, Day 8, 30 minutes |  |  |  |  |  | 0.0033 (0.00283) |  |
  CD4+CD25hiFoxP3+T cells, Day 8, 2 hours: number analyzed (Participants) | 0 | 14 | 0 | 17 | 0 | 0 | 6 | 4
  CD4+CD25hiFoxP3+T cells, Day 8, 2 hours |  | 0.0035 (0.00336) |  | 0.0015 (0.00265) |  |  | 0.0013 (0.00178) | 0.0055 (0.00466)
  CD4+CD25hiFoxP3+T cells, Day 8, 2.25 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0
  CD4+CD25hiFoxP3+T cells, Day 8, 2.25 hours |  |  |  |  | 0.0034 (0.00409) |  |  |
  CD4+CD25hiFoxP3+T cells, Day 8, 2.5 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
  CD4+CD25hiFoxP3+T cells, Day 8, 2.5 hours |  |  |  |  |  | 0.0027 (0.00293) |  |
  CD4+CD25hiFoxP3+T cells, Day 8, 4 hours: number analyzed (Participants) | 0 | 13 | 0 | 18 | 0 | 0 | 6 | 4
  CD4+CD25hiFoxP3+T cells, Day 8, 4 hours |  | 0.0038 (0.00380) |  | 0.0017 (0.00285) |  |  | 0.0012 (0.00125) | 0.0047 (0.00379)
  CD4+CD25hiFoxP3+T cells, Day 28: number analyzed (Participants) | 0 | 14 | 0 | 15 | 6 | 8 | 6 | 4
  CD4+CD25hiFoxP3+T cells, Day 28 |  | 0.0132 (0.01176) |  | 0.0096 (0.01231) | 0.0163 (0.00740) | 0.0200 (0.01421) | 0.0163 (0.00635) | 0.0253 (0.01205)
  CD8+CD25+FoxP3+T cells, Baseline: number analyzed (Participants) | 0 | 12 | 0 | 18 | 6 | 8 | 6 | 4
  CD8+CD25+FoxP3+T cells, Baseline |  | 0.0001 (0.00264) |  | 0.0032 (0.00699) | 0.0230 (0.03795) | -0.0086 (0.02386) | 0.0020 (0.00153) | 0.0027 (0.00825)
  CD8+CD25+FoxP3+T cells, Day 8, pre-dose |  | 0.0006 (0.00211) |  | 0.0011 (0.00302) | 0.0048 (0.01791) | 0.0054 (0.00563) | 0.0000 (0.00213) | -0.0006 (0.00360)
  CD8+CD25+FoxP3+T cells, Day 8, 15 minutes: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0
  CD8+CD25+FoxP3+T cells, Day 8, 15 minutes |  |  |  |  | 0.0096 (0.01322) |  |  |
  CD8+CD25+FoxP3+T cells, Day 8, 30 minutes: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
  CD8+CD25+FoxP3+T cells, Day 8, 30 minutes |  |  |  |  |  | 0.0138 (0.03663) |  |
  CD8+CD25+FoxP3+T cells, Day 8, 2 hours: number analyzed (Participants) | 0 | 14 | 0 | 17 | 0 | 0 | 6 | 4
  CD8+CD25+FoxP3+T cells, Day 8, 2 hours |  | 0.0020 (0.00241) |  | 0.0005 (0.00291) |  |  | -0.0001 (0.00187) | 0.0036 (0.00420)
  CD8+CD25+FoxP3+T cells, Day 8, 2.25 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0
  CD8+CD25+FoxP3+T cells, Day 8, 2.25 hours |  |  |  |  | -0.0057 (0.01376) |  |  |
  CD8+CD25+FoxP3+T cells, Day 8, 2.5 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
  CD8+CD25+FoxP3+T cells, Day 8, 2.5 hours |  |  |  |  |  | 0.0045 (0.01405) |  |
  CD8+CD25+FoxP3+T cells, Day 8, 4 hours: number analyzed (Participants) | 0 | 13 | 0 | 18 | 0 | 0 | 6 | 4
  CD8+CD25+FoxP3+T cells, Day 8, 4 hours |  | 0.0052 (0.01082) |  | -0.0006 (0.00443) |  |  | 0.0007 (0.00085) | 0.0008 (0.00459)
  CD8+CD25+FoxP3+T cells, Day 28: number analyzed (Participants) | 0 | 14 | 0 | 16 | 6 | 8 | 6 | 4
  CD8+CD25+FoxP3+T cells, Day 28 |  | 0.0036 (0.00443) |  | -0.0045 (0.01304) | 0.0037 (0.01012) | 0.0005 (0.01527) | 0.0004 (0.00382) | 0.0105 (0.01099)

12. Secondary Outcome: Mean Lymphocytes Subsets (CD4+ T Cells, CD8+ T Cells) Count
Description: One sample was collected at the screening visit and at Baseline. On dose Day 1, samples were collected at EOI and 4 hour post-SOI. On all other dosing days, samples were collected at pre-dose, EOI and 4 hour post-SOI. To obtain absolute counts for each lymphocyte subset (CD4+ T cells, CD8+ T cells) the proportion of total lymphocytes constituting that subset was multiplied by the total count for the same participant at the same time point. The data was collected on Baseline, Days 1 to 8, Days 14, 21, 28, Weeks 6, 8, 10, 12, Months 4, 5, 6, 12, 24, 36 and 48. However data for Days 8 and 28 is presented.
Time Frame: Day 8 and 28
Population: PD summary Population. Only those participants available at the specified time points were analyzed. Data for only quantifiable concentration is presented.
Measure: Mean (Standard Deviation); unit: Cells per microliter
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Number analyzed (Participants) | 0 | 14 | 17 | 18 | 7 | 9 | 6 | 4
Cells per microliter
  CD4+ T cells, Baseline: number analyzed (Participants) | 0 | 12 | 16 | 18 | 6 | 8 | 6 | 4
  CD4+ T cells, Baseline |  | 0.943 (0.2982) | 0.841 (0.2111) | 0.959 (0.2726) | 0.802 (0.1535) | 0.929 (0.1879) | 0.961 (0.5173) | 1.007 (0.2653)
  CD4+ T cells, Day 8: number analyzed (Participants) | 0 | 0 | 17 | 0 | 0 | 0 | 0 | 0
  CD4+ T cells, Day 8 |  |  | 0.636 (0.1741) |  |  |  |  |
  CD4+ T cells, Day 8, pre-dose: number analyzed (Participants) | 0 | 14 | 0 | 18 | 7 | 9 | 6 | 4
  CD4+ T cells, Day 8, pre-dose |  | 0.463 (0.1928) |  | 0.416 (0.1511) | 0.327 (0.1175) | 0.329 (0.1348) | 0.188 (0.0867) | 0.386 (0.1154)
  CD4+ T cells, Day 8, 15 minutes: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0
  CD4+ T cells, Day 8, 15 minutes |  |  |  |  | 0.233 (0.1504) |  |  |
  CD4+ T cells, Day 8, 30 minutes: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
  CD4+ T cells, Day 8, 30 minutes |  |  |  |  |  | 0.113 (0.0779) |  |
  CD4+ T cells, Day 8, 2 hours: number analyzed (Participants) | 0 | 14 | 0 | 17 | 0 | 0 | 6 | 4
  CD4+ T cells, Day 8, 2 hours |  | 0.296 (0.1341) |  | 0.210 (0.1781) |  |  | 0.108 (0.1202) | 0.099 (0.0553)
  CD4+ T cells, Day 8, 2.25 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0
  CD4+ T cells, Day 8, 2.25 hours |  |  |  |  | 0.218 (0.1569) |  |  |
  CD4+ T cells, Day 8, 2.5 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
  CD4+ T cells, Day 8, 2.5 hours |  |  |  |  |  | 0.117 (0.0502) |  |
  CD4+ T cells, Day 8, 4 hours: number analyzed (Participants) | 0 | 13 | 0 | 18 | 0 | 0 | 6 | 4
  CD4+ T cells, Day 8, 4 hours |  | 0.397 (0.1779) |  | 0.267 (0.1799) |  |  | 0.126 (0.0962) | 0.112 (0.0469)
  CD4+ T cells, Day 28: number analyzed (Participants) | 0 | 14 | 15 | 16 | 6 | 8 | 6 | 4
  CD4+ T cells, Day 28 |  | 0.835 (0.2971) | 0.812 (0.2211) | 0.978 (0.3193) | 0.743 (0.1846) | 0.797 (0.1824) | 0.927 (0.2153) | 0.689 (0.2199)
  CD8+ T cells, Baseline: number analyzed (Participants) | 0 | 12 | 16 | 18 | 6 | 8 | 6 | 4
  CD8+ T cells, Baseline |  | 0.586 (0.2370) | 0.442 (0.1404) | 0.425 (0.1213) | 0.466 (0.1720) | 0.519 (0.2813) | 0.437 (0.1761) | 0.638 (0.1711)
  CD8+ T cells, Day 8: number analyzed (Participants) | 0 | 0 | 17 | 0 | 0 | 0 | 0 | 0
  CD8+ T cells, Day 8 |  |  | 0.324 (0.1370) |  |  |  |  |
  CD8+ T cells, Day 8, pre-dose: number analyzed (Participants) | 0 | 14 | 0 | 18 | 7 | 9 | 6 | 4
  CD8+ T cells, Day 8, pre-dose |  | 0.242 (0.1133) |  | 0.192 (0.0873) | 0.149 (0.0297) | 0.161 (0.0815) | 0.143 (0.1248) | 0.298 (0.1108)
  CD8+ T cells, Day 8, 15 minutes: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0
  CD8+ T cells, Day 8, 15 minutes |  |  |  |  | 0.124 (0.0577) |  |  |
  CD8+ T cells, Day 8, 30 minutes: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
  CD8+ T cells, Day 8, 30 minutes |  |  |  |  |  | 0.093 (0.0558) |  |
  CD2+ T cells, Day 8, 2 hours: number analyzed (Participants) | 0 | 14 | 0 | 17 | 0 | 0 | 6 | 4
  CD2+ T cells, Day 8, 2 hours |  | 0.183 (0.1143) |  | 0.134 (0.0981) |  |  | 0.072 (0.0776) | 0.121 (0.0731)
  CD8+ T cells, Day 8, 2.25 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0
  CD8+ T cells, Day 8, 2.25 hours |  |  |  |  | 0.120 (0.0563) |  |  |
  CD8+ T cells, Day 8, 2.5 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
  CD8+ T cells, Day 8, 2.5 hours |  |  |  |  |  | 0.076 (0.0323) |  |
  CD8+ T cells, Day 8, 4 hours: number analyzed (Participants) | 0 | 13 | 0 | 18 | 0 | 0 | 6 | 4
  CD8+ T cells, Day 8, 4 hours |  | 0.211 (0.1255) |  | 0.150 (0.1013) |  |  | 0.095 (0.0857) | 0.138 (0.0313)
  CD8+ T cells, Day 28: number analyzed (Participants) | 0 | 14 | 15 | 16 | 6 | 8 | 6 | 4
  CD8+ T cells, Day 28 |  | 0.533 (0.1924) | 0.460 (0.1578) | 0.510 (0.2168) | 0.378 (0.0906) | 0.444 (0.1838) | 0.779 (0.3551) | 0.507 (0.1596)

13. Secondary Outcome: Mean CD4+/CD8+ Ratio
Description: One sample was collected at the screening visit and at Baseline. On dose Day 1, samples were collected at EOI and 4 hour post-SOI. On all other dosing days, samples were collected at pre-dose, EOI and 4 hour post-SOI. CD4+/CD8+ ratio was determined by dividing the absolute count of CD4+ T cells by the absolute count of CD8+ T cells for the same participant at the same time point. The data was collected on Baseline, Days 1 to 8, Days 14, 21, 28, Weeks 6, 8, 10, 12, Months 4, 5, 6, 12, 24, 36 and 48. However data for Days 8 and 28 is presented.
Time Frame: Day 8 and 28
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Number analyzed (Participants) | 0 | 14 | 17 | 18 | 7 | 9 | 6 | 4
Ratio
  Baseline: number analyzed (Participants) | 0 | 13 | 16 | 18 | 6 | 8 | 6 | 4
  Baseline |  | 1.95 (0.952) | 2.00 (0.551) | 2.35 (0.783) | 1.81 (0.339) | 2.14 (0.846) | 2.38 (1.099) | 1.64 (0.465)
  Day 8: number analyzed (Participants) | 0 | 0 | 17 | 0 | 0 | 0 | 0 | 0
  Day 8 |  |  | 2.12 (0.531) |  |  |  |  |
  Day 8, pre-dose: number analyzed (Participants) | 0 | 14 | 0 | 18 | 7 | 9 | 6 | 4
  Day 8, pre-dose |  | 2.15 (0.965) |  | 2.36 (0.958) | 2.15 (0.467) | 2.12 (0.564) | 1.80 (0.932) | 1.34 (0.276)
  Day 8, 15 minutes: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0
  Day 8, 15 minutes |  |  |  |  | 1.72 (0.684) |  |  |
  Day 8, 30 minutes: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
  Day 8, 30 minutes |  |  |  |  |  | 1.17 (0.547) |  |
  Day 8, 2 hours: number analyzed (Participants) | 0 | 14 | 0 | 18 | 0 | 0 | 6 | 4
  Day 8, 2 hours |  | 1.82 (0.740) |  | 1.51 (0.728) |  |  | 1.62 (1.163) | 0.85 (0.255)
  Day 8, 2.25 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0
  Day 8, 2.25 hours |  |  |  |  | 1.72 (0.731) |  |  |
  Day 8, 2.5 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
  Day 8, 2.5 hours |  |  |  |  |  | 1.56 (0.441) |  |
  Day 8, 4 hours: number analyzed (Participants) | 0 | 14 | 0 | 18 | 0 | 0 | 6 | 4
  Day 8, 4 hours |  | 2.11 (0.906) |  | 1.86 (0.873) |  |  | 1.72 (1.079) | 0.80 (0.239)
  Day 8, 10 hours: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Day 8, 10 hours |  | 1.36 (NA) — Only one participant was analyzed, hence no data. |  |  |  |  |  |
  Day 28: number analyzed (Participants) | 0 | 14 | 16 | 16 | 6 | 8 | 6 | 4
  Day 28 |  | 1.69 (0.684) | 1.87 (0.339) | 2.08 (0.838) | 2.00 (0.357) | 2.02 (0.829) | 1.61 (1.263) | 1.38 (0.319)

14. Secondary Outcome: Percent Lymphocytes Subsets (CD25+CD8+Tregs) Count
Description: One sample was collected at the screening visit and at Baseline. On dose Day 1, samples were collected at EOI and 4 hour post-SOI. On all other dosing days, samples were collected at pre-dose, EOI and 4 hour post-SOI. The data was collected on Baseline, Days 1 to 8, Days 14, 21, 28, Weeks 6, 8, 10, 12, Months 4, 5, 6, 12, 24, 36 and 48. However data for Days 8 and 28 is presented.
Time Frame: Day 8 and 28
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percentage of lymphocytes
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Number analyzed (Participants) | 0 | 0 | 17 | 0 | 0 | 0 | 0 | 0
Percentage of lymphocytes
  Baseline: number analyzed (Participants) | 0 | 0 | 16 | 0 | 0 | 0 | 0 | 0
  Baseline |  |  | 20.71 (25.324) |  |  |  |  |
  Day 8 |  |  | 22.08 (23.486) |  |  |  |  |
  Day 28: number analyzed (Participants) | 0 | 0 | 16 | 0 | 0 | 0 | 0 | 0
  Day 28 |  |  | 35.62 (28.538) |  |  |  |  |

15. Secondary Outcome: Amounts of Cell-bound Otelixizumab on CD4+ and CD8+ T Cells
Description: Samples were planned to analyze at the screening visit and at Baseline. Further on dose Day 1, at EOI and 4 hour post-SOI. On all other dosing days, at pre-dose, EOI and 4 hour post-SOI up to 48 months.
Time Frame: At the screening visit and at Baseline. On dose Day 1, at EOI and 4 hour post-SOI. On all other dosing days, at pre-dose, EOI and 4 hour post-SOI up to 48 months.
Population: PD summary Population. Data was not collected for this endpoint.
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Saturation of CD4+ and CD8+ T Cells With Otelixizumab
Description: as for outcome 15
Time Frame: as for outcome 15
Population: PD summary Population. Data was not collected for this endpoint.
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: CD3/TCR Complexes on CD4+ and CD8+ T Cells
Description: Samples were planned to analyze at the Screen visit and at Baseline. Further on dose Day 1, at EOI and 4 hour post-SOI. On all other dosing days, at pre-dose, EOI and 4 hour post-SOI up to 48 months.
Time Frame: At the Screen visit and at Baseline. On dose Day 1, at EOI and 4 hour post-SOI. On all other dosing days, at pre-dose, EOI and 4 hour post-SOI up to 48 months.
Population: PD summary Population. Data was not collected for this endpoint.
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Detectable Anti-otelixizumab Antiglobulin Response
Description: Anti-otelixizumab antibody levels were determined by ELISA. Immunogenicity data was not collected for Cohort 5 (5 day dosing) participants.
Time Frame: Up to Month 48
Population: All subjects Population. Participants from all 7 cohorts who had received a total dose <3.0 mg were analyzed as a separate treatment group. Immunogenicity data was not collected for Cohort 5 (5 day dosing) participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Number analyzed (Participants) | 8 | 15 | 0 | 19 | 7 | 9 | 6 | 6
Participants | 0 | 0 |  | 1 | 0 | 0 | 2 | 0

19. Secondary Outcome: Number of Participants With Use of Analgesics, Antihistamines and IV Hydration as Concomitant Medication During Dosing Days
Description: Ibuprofen (analgesic) was given orally as follows: 400-800 mg 2 hour before SOI, 400-800 mg 2 hour after SOI, 400-800 mg 6 hour after SOI, and 400-800 mg at bedtime. If ibuprofen was contraindicated, acetaminophen was used in place of ibuprofen. Acetaminophen doses were adjusted so as it did not exceed 1000 mg per 6 hour or 4000 mg per day. A non-sedating antihistamine (cetirizine) was administered approximately 1 hour prior to each infusion of study drug. The recommended initial dose of cetirizine was 5 mg or 10 mg per day in adults and children aged 12 years and older. Normal saline solution was administered IV as needed to maintain hydration.
Time Frame: Up to Day 8
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Number analyzed (Participants) | 8 | 15 | 18 | 19 | 7 | 9 | 6 | 6
Participants
  Day 1, Analgesics | 8 | 11 | 18 | 19 | 4 | 6 | 3 | 6
  Day 1, Antihistamines | 8 | 11 | 18 | 19 | 4 | 6 | 3 | 6
  Day 1, IV Saline | 6 | 13 | 13 | 16 | 3 | 3 | 3 | 5
  Day 2, Analgesics | 8 | 11 | 17 | 19 | 4 | 6 | 3 | 6
  Day 2, Antihistamines | 8 | 11 | 18 | 19 | 4 | 6 | 3 | 6
  Day 2, IV Saline | 7 | 13 | 14 | 18 | 4 | 2 | 3 | 5
  Day 3, Analgesics: number analyzed (Participants) | 7 | 15 | 18 | 19 | 7 | 9 | 6 | 6
  Day 3, Analgesics | 7 | 11 | 18 | 19 | 4 | 6 | 3 | 6
  Day 3, Antihistamines: number analyzed (Participants) | 7 | 15 | 18 | 19 | 7 | 9 | 6 | 6
  Day 3, Antihistamines | 7 | 11 | 18 | 19 | 4 | 6 | 3 | 6
  Day 3, IV Saline: number analyzed (Participants) | 7 | 15 | 18 | 19 | 7 | 9 | 6 | 6
  Day 3, IV Saline | 6 | 13 | 14 | 17 | 4 | 3 | 3 | 5
  Day 4, Analgesics: number analyzed (Participants) | 5 | 15 | 18 | 19 | 7 | 9 | 6 | 6
  Day 4, Analgesics | 5 | 11 | 18 | 19 | 4 | 6 | 3 | 6
  Day 4, Antihistamines: number analyzed (Participants) | 5 | 15 | 18 | 19 | 7 | 9 | 6 | 6
  Day 4, Antihistamines | 5 | 11 | 18 | 19 | 4 | 6 | 3 | 6
  Day 4, IV Saline: number analyzed (Participants) | 5 | 15 | 18 | 19 | 7 | 9 | 6 | 6
  Day 4, IV Saline | 5 | 13 | 14 | 17 | 4 | 4 | 3 | 6
  Day 5, Analgesics: number analyzed (Participants) | 2 | 15 | 18 | 19 | 7 | 9 | 6 | 6
  Day 5, Analgesics | 2 | 11 | 17 | 19 | 4 | 6 | 3 | 6
  Day 5, Antihistamines: number analyzed (Participants) | 2 | 15 | 18 | 19 | 7 | 9 | 6 | 6
  Day 5, Antihistamines | 2 | 11 | 17 | 18 | 4 | 6 | 3 | 6
  Day 5, IV Saline: number analyzed (Participants) | 2 | 15 | 18 | 19 | 7 | 9 | 6 | 6
  Day 5, IV Saline | 2 | 13 | 14 | 17 | 4 | 5 | 2 | 6
  Day 6, Analgesics: number analyzed (Participants) | 1 | 15 | 0 | 19 | 7 | 9 | 6 | 6
  Day 6, Analgesics | 1 | 15 |  | 19 | 4 | 6 | 3 | 6
  Day 6, Antihistamines: number analyzed (Participants) | 1 | 15 | 0 | 19 | 7 | 9 | 6 | 6
  Day 6, Antihistamines | 1 | 11 |  | 19 | 4 | 6 | 3 | 6
  Day 6, IV Saline: number analyzed (Participants) | 8 | 15 | 0 | 19 | 7 | 9 | 6 | 6
  Day 6, IV Saline | 0 | 13 |  | 17 | 4 | 3 | 2 | 6
  Day 7, Analgesics: number analyzed (Participants) | 0 | 15 | 0 | 19 | 7 | 9 | 6 | 6
  Day 7, Analgesics |  | 11 |  | 19 | 4 | 6 | 3 | 6
  Day 7, Antihistamines: number analyzed (Participants) | 0 | 15 | 0 | 19 | 7 | 9 | 6 | 6
  Day 7, Antihistamines |  | 11 |  | 19 | 3 | 6 | 3 | 6
  Day 7, IV Saline: number analyzed (Participants) | 0 | 15 | 0 | 19 | 7 | 9 | 6 | 6
  Day 7, IV Saline |  | 14 |  | 18 | 4 | 3 | 3 | 6
  Day 8, Analgesics: number analyzed (Participants) | 0 | 15 | 0 | 19 | 7 | 9 | 6 | 5
  Day 8, Analgesics |  | 12 |  | 18 | 4 | 6 | 3 | 5
  Day 8, Antihistamines: number analyzed (Participants) | 0 | 15 | 0 | 19 | 7 | 9 | 6 | 5
  Day 8, Antihistamines |  | 12 |  | 19 | 4 | 5 | 2 | 5
  Day 8, IV Saline: number analyzed (Participants) | 0 | 15 | 0 | 19 | 7 | 9 | 6 | 5
  Day 8, IV Saline |  | 14 |  | 18 | 4 | 3 | 3 | 5

20. Secondary Outcome: Change From Baseline in Percent Glycosylated Hemoglobin (HbA1c)
Description: Participants were seen weekly during the first 4 weeks post-dose and then every other week through Week 12. After Week 12, visits occurred every 1 to 3 months through Month 18, which completes the Core Study up to Month 48 (follow up). Day 1 pre-dose value was considered as Baseline value. Change from Baseline was post-Baseline value minus Baseline value.
Time Frame: Baseline and up to Month 48
Population: PD summary Population. Only those participants available at the specified time points were analyzed. Participants from all 7 cohorts who had received a total dose <3.0 mg were analyzed as a separate treatment group. Data for only quantifiable concentration is presented.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
Number analyzed (Participants) | 0 | 14 | 17 | 18 | 7 | 9 | 6 | 4
Percentage of glycosylated hemoglobin
  Day 28: number analyzed (Participants) | 0 | 13 | 16 | 17 | 5 | 7 | 6 | 4
  Day 28 |  | -0.58 (0.656) | -0.44 (0.788) | -0.41 (0.404) | -0.44 (0.416) | -0.60 (0.624) | -0.88 (0.578) | -0.53 (0.737)
  Week 6: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Week 6 |  |  |  | 0.10 (NA) — Only one participant was analyzed, hence no data. |  |  | -0.20 (NA) — Only one participant was analyzed, hence no data. |
  Week 8: number analyzed (Participants) | 0 | 13 | 16 | 17 | 6 | 8 | 6 | 4
  Week 8 |  | -0.69 (0.825) | -0.48 (1.187) | -0.19 (0.749) | -0.48 (0.618) | -0.64 (0.838) | -0.90 (1.277) | -0.72 (1.124)
  Week 10: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Week 10 |  |  |  | -0.10 (NA) — Only one participant was analyzed, hence no data. |  |  |  |
  Week 12: number analyzed (Participants) | 0 | 13 | 16 | 17 | 6 | 7 | 6 | 4
  Week 12 |  | -0.35 (0.670) | -0.15 (1.272) | 0.19 (0.534) | -0.37 (0.784) | -0.64 (1.180) | -0.55 (1.063) | -0.30 (1.494)
  Month 4: number analyzed (Participants) | 0 | 12 | 14 | 16 | 6 | 7 | 6 | 4
  Month 4 |  | 0.08 (0.890) | 0.35 (1.575) | 0.39 (0.545) | -0.18 (1.061) | 0.39 (1.497) | -0.17 (1.124) | 0.05 (1.196)
  Month 5: number analyzed (Participants) | 0 | 12 | 15 | 17 | 6 | 6 | 6 | 4
  Month 5 |  | 0.10 (0.867) | 0.76 (1.790) | 0.42 (0.797) | 0.13 (0.999) | 0.63 (1.435) | -0.07 (0.983) | 0.55 (1.338)
  Month 6: number analyzed (Participants) | 0 | 12 | 15 | 17 | 5 | 7 | 6 | 4
  Month 6 |  | -0.23 (0.819) | 0.43 (1.479) | 0.22 (1.274) | -0.28 (0.743) | 0.61 (1.655) | -0.25 (0.985) | 0.00 (1.699)
  Month 9: number analyzed (Participants) | 0 | 12 | 15 | 17 | 6 | 7 | 5 | 4
  Month 9 |  | -0.43 (0.878) | 1.03 (1.589) | 0.26 (1.118) | 0.10 (1.307) | 0.19 (1.558) | -0.64 (1.076) | -0.00 (2.304)
  Month 12: number analyzed (Participants) | 0 | 10 | 12 | 17 | 5 | 6 | 6 | 4
  Month 12 |  | -0.27 (0.800) | 1.31 (1.729) | 0.36 (1.330) | 0.90 (1.938) | 0.90 (2.045) | -0.23 (0.784) | 0.35 (2.412)
  Month 16: number analyzed (Participants) | 0 | 9 | 9 | 14 | 6 | 7 | 5 | 3
  Month 16 |  | -0.36 (0.886) | 0.93 (1.542) | 0.45 (1.591) | 0.20 (1.284) | 1.33 (2.368) | 0.06 (0.573) | 0.00 (2.358)
  Month 18: number analyzed (Participants) | 0 | 9 | 4 | 13 | 6 | 7 | 6 | 4
  Month 18 |  | -0.24 (1.184) | 0.27 (1.087) | 0.58 (1.476) | 0.15 (1.323) | 1.06 (2.277) | -0.33 (1.253) | 0.42 (2.138)
  Month 24: number analyzed (Participants) | 0 | 10 | 0 | 12 | 6 | 7 | 6 | 3
  Month 24 |  | -0.32 (1.172) |  | 0.31 (1.059) | 0.38 (1.714) | 1.66 (3.730) | -0.25 (1.141) | 0.20 (2.117)
  Month 36: number analyzed (Participants) | 0 | 8 | 0 | 10 | 1 | 6 | 6 | 0
  Month 36 |  | -0.21 (1.212) |  | 0.85 (1.090) | -0.10 (NA) — Only one participant was analyzed, hence no data. | 2.03 (3.063) | -0.55 (1.677) |
  Month 48: number analyzed (Participants) | 0 | 7 | 0 | 4 | 0 | 0 | 0 | 0
  Month 48 |  | -0.24 (0.648) |  | 0.20 (1.254) |  |  |  |

ADVERSE EVENTS:
Time Frame: All SAEs and non-SAEs were collected up to Month 24
Description: SAEs and non-SAEs were reported for All subjects Population. Participants from all 7 cohorts who had received a total dose <3.0 mg were analyzed as a separate treatment group. All other participants were analyzed according to the planned dose based on the cohort they belonged to.
Arm/Group | Otelixizumab <3.0 mg | Otelixizumab 3.1 mg | Otelixizumab 3.1 mg (5 Days) | Otelixizumab 4.35 mg | Otelixizumab 4.35 mg (ITC-15) | Otelixizumab 4.35 mg (ITC-30) | Otelixizumab 6.85 mg | Otelixizumab 8.85 mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/15 | 0/18 | 0/19 | 0/7 | 0/9 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/8 | 2/15 | 1/18 | 0/19 | 0/7 | 1/9 | 1/6 | 2/6
Other Adverse Events (participants affected / at risk) | 8/8 | 15/15 | 18/18 | 18/19 | 7/7 | 9/9 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Otelixizumab <3.0 mg (N=8) | Otelixizumab 3.1 mg (N=15) | Otelixizumab 3.1 mg (5 Days) (N=18) | Otelixizumab 4.35 mg (N=19) | Otelixizumab 4.35 mg (ITC-15) (N=7) | Otelixizumab 4.35 mg (ITC-30) (N=9) | Otelixizumab 6.85 mg (N=6) | Otelixizumab 8.85 mg (N=6)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis enteroviral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Otelixizumab <3.0 mg (N=8) | Otelixizumab 3.1 mg (N=15) | Otelixizumab 3.1 mg (5 Days) (N=18) | Otelixizumab 4.35 mg (N=19) | Otelixizumab 4.35 mg (ITC-15) (N=7) | Otelixizumab 4.35 mg (ITC-30) (N=9) | Otelixizumab 6.85 mg (N=6) | Otelixizumab 8.85 mg (N=6)
Headache (Nervous system disorders) | 8 | 12 | 18 | 18 | 7 | 9 | 6 | 6
Dizziness (Nervous system disorders) | 1 | 1 | 3 | 5 | 0 | 1 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neurological symptom (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 3 | 5 | 7 | 5 | 2 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 2 | 5 | 0 | 2 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 3 | 2 | 3 | 1 | 0 | 2 | 1
Influenza (Infections and infestations) | 1 | 1 | 2 | 1 | 0 | 2 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 2 | 1 | 1 | 0 | 2 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion site cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lice infestation (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 6 | 9 | 9 | 14 | 4 | 4 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight fluctuation (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 3 | 11 | 10 | 3 | 1 | 5 | 2
Vomiting (Gastrointestinal disorders) | 4 | 2 | 7 | 3 | 2 | 0 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 4 | 2 | 1 | 1 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 4 | 0 | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 3 | 1 | 5 | 6 | 2 | 1 | 4 | 2
Pyrexia (General disorders) | 1 | 3 | 4 | 3 | 2 | 1 | 2 | 3
Fatigue (General disorders) | 1 | 3 | 3 | 2 | 0 | 2 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Infusion site phlebitis (General disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Infusion site erythema (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Catheter site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site rash (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion site induration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion site scab (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pitting oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sensation of foreign body (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 6 | 3 | 0 | 3 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 3 | 0 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 3 | 1 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 2 | 0 | 2 | 1
Rash maculo-papular (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Circumoral oedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermographism (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin striae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 3 | 1 | 3 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 2 | 2 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 3 | 1 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngeal lesion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 2 | 1 | 3 | 2 | 0 | 3 | 1
Hypotension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 2
Hypertension (Vascular disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 1 | 4 | 1 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 0 | 5 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Platelet disorder (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chemical eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid pain (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Blood iron decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Epstein-Barr virus test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hormone level abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Balanitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast calcifications (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
This study was terminated on 15 December 2011

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.